CLINICAL TRIAL: NCT05361837
Title: Efficacy of Single Level Versus Bilevel Serratus Anterior Plane Block With Dexmedetomidine During Breast Cancer Surgery
Brief Title: Efficacy of Serratus Anterior Plane Block With Dexmedetomidine During Breast Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AP2204-50104
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single level serratus anterior plane block (Active Comparator): the allocated patients will receive single injection serratus anterior plane block at the level of third rib with local anesthetics only
  Interventions: Procedure: Single level serratus anterior plane block
- Single level serratus anterior plane block with dexmedetomidine (Experimental): the allocated patients will receive single injection serratus anterior plane block at the level of third rib with local anesthetics and dexmedetomidine
  Interventions: Procedure: Single level serratus anterior plane block with dexmedetomidine
- Bilevel serratus anterior plane block (Experimental): the allocated patients will receive injection serratus anterior plane block at 2 levels, the level of third rib and the level of the fifth rib with local anesthetics only
  Interventions: Procedure: Bilevel serratus anterior plane block
- Bilevel serratus anterior plane block with dexmedetomidine (Experimental): the allocated patients will receive injection serratus anterior plane block at 2 levels, the level of third rib and the level of the fifth rib with local anesthetics and dexmedetomidine
  Interventions: Procedure: Bilevel serratus anterior plane block with dexmedetomidine

INTERVENTIONS:
Procedure: Single level serratus anterior plane block — Serratus anterior plane block with local anesthetics at the third rib
  Arms: Single level serratus anterior plane block
Procedure: Single level serratus anterior plane block with dexmedetomidine — Serratus anterior plane block with local anesthetics and dexmedetomidine at the third rib
  Arms: Single level serratus anterior plane block with dexmedetomidine
Procedure: Bilevel serratus anterior plane block — Serratus anterior plane block with local anesthetics at the third and fifth rib
  Arms: Bilevel serratus anterior plane block
Procedure: Bilevel serratus anterior plane block with dexmedetomidine — Serratus anterior plane block with local anesthetics and dexmedetomidine at the third and fifth rib
  Arms: Bilevel serratus anterior plane block with dexmedetomidine

SUMMARY:
This study aims to compare single level serratus block versus bilevel serratus block with and without dexmedetomidine in cancer patients undergoing modified radical mastectomy for breast cancer regarding pain control and possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for modified radical mastectomy,
* Age 18-65 years,
* ASA I-II

Exclusion Criteria:

* patient refusal,
* coagulation defects,
* abnormal kidney or liver functions,
* local infection at site of injection.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 172 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
First time to receive analgesia | First 24 hours postoperatively
  first time to receive morphine analgesia in hours
Total analgesic requisite | First 24 hours postoperatively
  total amount of morphine consumption in the first 24 hours postoperatively in mg

SECONDARY OUTCOMES:
Pain scores | First 24 hours postoperatively
  pain scores will be assessed using Visual Analogue Scale on a sale from 0 to 10 with 0 meanung no pain and 10 meaning severe pain
Side effects | First 24 hours postoperatively
  nausea and vomiting and hematoma at site of injection
Perioperative heart rate values | First 24 hours
  heart rate values in the form of beat per minute in the perioperative period including preoperative, intraoperative and postoperative
Mean arterial blood pressure | First 24 hours
  Mean arterial blood pressure values in the form mmHg in the perioperative period including preoperative, intraoperative and postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant Professor of Anesthesia and Pain management
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided